CLINICAL TRIAL: NCT05668585
Title: A Phase 1/2 Open-Label Multicenter Trial to Characterize the Safety, Tolerability, and Preliminary Efficacy of CFT1946 as Monotherapy and Combination Therapy in Subjects With BRAF V600 Mutant Solid Tumors
Brief Title: A Study to Characterize the Safety, Tolerability, and Preliminary Efficacy of CFT1946 as Monotherapy and Combination Therapy in Subjects With BRAF V600 Mutant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C4 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFT1946-1101
Record Dates: First submitted 2022-12-06; First posted 2022-12-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors; Melanoma; NSCLC; CRC; ATC
Keywords: Solid Tumors; Melanoma; NSCLC; ATC; BRAF mutant; CRC
MeSH Terms: conditions — Melanoma | interventions — trametinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1: Arm A: CFT1946 (Experimental): Approximately 40 subjects with V600 Solid Tumors (non-CNS) (post BRAF inhibitor for NSCLC, CRC, melanoma, ATC)
  Interventions: Drug: CFT1946
- Phase 1: Arm B: CFT1946 + trametinib (Experimental): Approximately 28 subjects with V600 Solid Tumors (non-CNS) (post BRAF inhibitor for NSCLC, CRC, melanoma)
  Interventions: Drug: CFT1946; Drug: Trametinib
- Phase 2: Arm A1: CFT1946 (Experimental): Approximately 30 subjects with V600 melanoma or NSCLC (post BRAF inhibitor)
  Interventions: Drug: CFT1946
- Phase 2: Arm B1: CFT1946 + trametinib (Experimental): Approximately 20 subjects with V600 melanoma or NSCLC (post BRAF Inhibitor)
  Interventions: Drug: CFT1946; Drug: Trametinib
- Phase 1: Arm C: CFT1946 + cetuximab (Experimental): Approximately 30 subjects with CRC (post BRAF inhibitor)
  Interventions: Drug: CFT1946; Drug: Cetuximab
- Phase 2: Arm C1: CFT1946 + cetuximab (Experimental): Approximately 40 subjects with CRC (post BRAF inhibitor)
  Interventions: Drug: CFT1946; Drug: Cetuximab

INTERVENTIONS:
Drug: CFT1946 — Specified oral dose on specified day
Drug: Trametinib — Specified oral dose on specified day
  Arms: Phase 1: Arm B: CFT1946 + trametinib; Phase 2: Arm B1: CFT1946 + trametinib
Drug: Cetuximab — Specified intravenous dose on specified day
  Arms: Phase 1: Arm C: CFT1946 + cetuximab; Phase 2: Arm C1: CFT1946 + cetuximab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of CFT1946 as well as to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of CFT1946 as monotherapy (Arm A) and in combination with trametinib (CFT1946 + trametinib; Arm B) or Cetuximab (CFT1946 + cetuximab; Arm C).

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative, where applicable) is willing and able to provide signed informed consent and can follow protocol requirements
2. Subject is ≥18 years of age at time of informed consent
3. Eastern Cooperative Oncology Group performance status of 0 or 1
4. Subject has documented evidence of a BRAF V600 mutation obtained from tumor tissue or liquid biopsy: (other protocol conditions may apply)
5. Subject must have received ≥1 prior line of SoC therapy for their unresectable locally advanced or metastatic disease with disease progression on or after last prior treatment. Prior regimens for these subjects vary by indication and investigational arm, but must have included the following:

   1. Melanoma or NSCLC (Phase 1 and Phase 2 Arms A1 and B1): Prior receipt of a BRAF inhibitor and an immune checkpoint inhibitor (any sequence or combination). Prior (neo)adjuvant immunotherapy may be acceptable.
   2. CRC: Subjects must have received no more than 4 lines of prior therapy which includes systemic chemotherapy-based regimen per SoC for unresectable locally advanced or metastatic disease, and previous treatment with BRAF inhibitor in combination with an EGFR monoclonal antibody. Subjects with documented MSI-H or dMMR CRC must have received prior immunotherapy. Subjects with MSS disease must have received at least 2 prior treatments. Subjects who received neo(adjuvant) chemotherapy regimens may be eligible.
   3. ATC: Subjects must have received SoC therapy options including BRAF inhibitor if available and of benefit to the subject
   4. Other BRAF V600 mutant solid tumors (non-CNS): Subjects must have received SoC therapy options per their Investigator's best judgment, including BRAF inhibitor if available and of benefit to the subject
6. Subject has measurable disease per RECIST v1.1
7. Adequate bone marrow, liver, renal, and cardiac function
8. A female subject may be eligible if not pregnant, planning a pregnancy, not breast feeding, a women of non-child bearing potential or a WOCBP willing to comply with protocol conditions relating to the use contraception, ova or blood donation and pregnancy testing prior to the first dose
9. A male subject must agree to comply with protocol conditions relating to the use of contraception, sperm and blood donation
10. Subject can safely swallow a tablet or pill

Other protocol defined exclusion criteria may apply

Exclusion Criteria:

1. Subject has had major surgery within 21 days prior to the planned first dose. Minor surgery is permitted within 21 days prior to enrollment
2. Subject with CNS involvement (primary tumor or metastatic disease), except if clinically stable, have no evidence of new or enlarging brain metastases and are on stable or tapering doses of steroids for at least 7 days prior to first dose. Subjects with untreated brain metastases may be eligible to enter without prior radiation therapy.
3. Subject with known malignancy other than trial indication that is progressing or has required treatment within the past 3 years, except for conditions that have undergone potentially curative therapy
4. Subject with history of thromboembolic or cerebrovascular events ≤6 months as defined in the protocol
5. Subject with impaired cardiac function or clinically significant cardiac disease, as defined in the protocol
6. Subject with history of uncontrolled diabetes mellitus (only for subjects who will receive CFT1946 + trametinib)
7. Subject with history or current evidence of retinal vein occlusion (RVO), chorioretinopathy, or current risk factors for RVO (only for subjects who will receive CFT1946 + trametinib)
8. Subject has received live, attenuated vaccine within 28 days prior to first dose administration
9. Subject has history of pneumonitis or interstitial lung disease
10. Subject has history of uveitis
11. Subject has clinically significant gastrointestinal abnormalities.
12. Subject has known human immunodeficiency virus (HIV) infection (with exceptions)
13. Subject has history of or known HBV or active HCV infection
14. Subject has concurrent administration of strong CYP3A4/5 inhibitors and inducers, including any herbal medications/supplements
15. Subject has presence of Grade ≥2 toxicity due to prior cancer therapy, excepting alopecia and hypothyroidism requiring thyroid replacement therapy
16. Subject has initiation or receipt of the following ≤7 days prior to first dose administration: Hematopoietic colony-stimulating growth factors, transfusion of packed red blood cells (pRBC), and transfusion of platelets
17. Subject is pregnant, breastfeeding, or expecting to conceive or father children any time during the study

Other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs and SAEs | From enrollment until 30 days after completion of study treatment
  Phase 1
Incidence of dose limiting toxicities (DLTs) | From enrollment until 28 days after first dose
  Phase 1
Number of subjects with changes between baseline and post-baseline safety assessments based on safety laboratory results graded by CTCAE v5.0 | From enrollment until 30 days after completion of study treatment
  Phase 1
Frequency of dose interruptions and dose reductions | From enrollment until 30 days after completion of study treatment
  Phase 1
Frequency of AEs leading to discontinuation of study treatment(s) | From enrollment until 30 days after completion of study treatment
  Phase 1
Overall response rate (ORR) | Up to approximately 43 months
  Phase 2 only according to RECIST v1.1 criteria
Disease control rate (DCR) at 3, 6, and 12 months | Up to 12 months
  Phase 2
Duration of Response (DOR) | Up to approximately 43 months
  Phase 2

SECONDARY OUTCOMES:
Frequency and severity of AEs and SAEs | From enrollment until 30 days after completion of study treatment
  Phase 2
Number of subjects with changes between baseline and post-baseline safety assessments based on safety laboratory results graded by CTCAE v5.0 | From enrollment until 30 days after completion of study treatment
  Phase 2
Frequency of dose interruptions and dose reductions | From enrollment until 30 days after completion of study treatment
  Phase 2
Frequency of AEs leading to discontinuation of study treatment(s) | From enrollment until 30 days after completion of study treatment
  Phase 2
Plasma concentration of CFT1946 to characterize the pharmacokinetics (PK) parameters of CFT1946 monotherapy and in combination with trametinib | Up to approximately 20 weeks
  Phase 1 and Phase 2
PK-QTcF relationship | Up to approximately 8 weeks
  Phase 1 and Phase 2
Overall response rate (ORR) | Up to approximately 43 months
  Phase 1
Disease control rate (DCR) at 3, 6, and 12 months | Up to 12 months
  Phase 1
Progression-free survival (PFS) | Up to approximately 43 months
  Phase 1 and Phase 2
Duration of response (DOR) | Up to approximately 43 months
  Phase 1
Assess the pharmacodynamics by percent reduction from baseline of target protein | At multiple time points up to 4 weeks
  Tumor BRAF-V600 degradation at scheduled timepoints

CONTACTS AND LOCATIONS:
Locations (26):
- United States (11):
  - University of Arizona - Cancer Center, Tucson, Arizona
  - Florida Cancer Specialists, Sarasota, Florida
  - Community Health Network, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Allina Health System DBA Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists (NEXT Oncology Virginia), Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- France (4):
  - Institut Bergonie, Bordeaux
  - Chu de Lille, Lille
  - Centre Leon Berard, Lyon
  - IUCT Oncopole, Toulouse
- Germany (2):
  - KEM | Evang. Kliniken Essen-Mitte gGmbH, Essen
  - Universitaetsklinikum Essen, Essen
- Spain (7):
  - NEXT Oncology Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jiminez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No